CLINICAL TRIAL: NCT03615885
Title: Acute Cardio-metabolic Responses to Different Forms of Montmorency Tart Cherry Supplementation in Humans With Metabolic Syndrome
Brief Title: Acute Cardio-metabolic Responses to Montmorency Tart Cherry Supplementation in Metabolic Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hertfordshire (Other)
Collaborators: Heart UK (Unknown)
Responsible Party: Principal Investigator, Terun Desai, PhD Student, University of Hertfordshire
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: LMS/PGT/UH/02843
Record Dates: First submitted 2018-07-20; First posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-07

CONDITIONS: Metabolic Syndrome; Insulin Resistance; Hypertension
Keywords: Montmorency Tart Cherry; Anthocyanins; Polyphenols; Metabolic Syndrome; Insulin Resistance; Hypertension; Lipid Profile
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo Drink (Placebo Comparator): Placebo drink attempted to match for total energy, appearance and taste of Montmorency tart cherry juice.
  Interventions: Dietary Supplement: Placebo
- Montmorency Tart Cherry Capsules (Experimental): 10 capsules consumed to match total anthocyanin content to Montmorency tart cherry juice.
  Interventions: Dietary Supplement: Montmorency Tart Cherry Capsules
- Montmorency Tart Cherry Juice (Experimental): Single-bolus of Montmorency tart cherry juice (130 mL)
  Interventions: Dietary Supplement: Montmorency Tart Cherry Juice

INTERVENTIONS:
Dietary Supplement: Montmorency Tart Cherry Capsules — Capsules are made from 100% natural, tart Montmorency cherries. Carefully prepared Montmorency cherry skins are freeze-dried and milled into a fine powder to protect the cherry phytonutrients and optimise absorbtion. This powder is then encapsulated into a 100% vegetarian shell.
  Arms: Montmorency Tart Cherry Capsules
Dietary Supplement: Montmorency Tart Cherry Juice — 100% natural, tart Montmorency cherry concentrate (30mL) diluted with 100mL water.
  Concentrate contains no sweeteners, preservatives, flavourings or added sugar.
  Arms: Montmorency Tart Cherry Juice
Dietary Supplement: Placebo — 130ml serving
  Placebo composition: Water (100ml), Cherry Cordial Concentrate (30ml), Citric Acid (1.5g), Maltodextrin (24.75g), Black Food Colouring (2ml).
  Arms: Placebo Drink

SUMMARY:
The present study examined the effect of Montmorency tart cherry juice and capsules on functional and blood-based cardio-metabolic markers in humans with Metabolic Syndrome. Participants received a single bolus of Montmorency tart cherry juice, Montmorency tart cherry capsules and placebo in a random, crossover trial. Outcome variables were measured immediately pre- and up to 5 hours post-bolus. It was hypothesised that Montmorency tart cherry juice and capsules would improve cardio-metabolic markers. Furthermore, it was hypothesised that Montmorency tart cherry capsules would be more beneficial than Montmorency tart cherry juice due to increased bioavailability of phytochemicals.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker,

Meet 3 of 5 criteria for Metabolic Syndrome based on National Cholesterol Education Program-Adult Treatment Panel III guidelines:

1. Waist Circumference: >102cm (men), >88cm (women)
2. Fasting Serum Triglycerides: ≥1.69 mmol.L-1
3. Fasting High Density Lipoprotein: <1.03 mmol.L-1 (men), <1.29 mmol.L-1 (women)
4. Blood Pressure: ≥130 mmHg SBP or ≥85 mmHg DBP
5. Fasting Plasma Glucose: ≥6.1 mmol.L-1

Exclusion Criteria:

* Current or previous history of gastrointestinal, cardiovascular, hepatic or renal disease, currently diagnosed with diabetes or uncontrolled hypertension (≥160/100 mmHg), allergy to maltodextrin or specific fruit products and those currently taking medication (such as steroids, NSAIDs, antibiotics, antihypertensive, hypoglycaemic, lipid-lowering drugs) or currently using any nutritional or antioxidant supplement. Heavy alcohol consumption (>14 units per week).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Fasting Insulin | Pre-Bolus and Post-Bolus (1hr, 3hr, 5hr)
Change in Fasting Lipid Profile (Total Cholesterol, HDL, Triglycerides, LDL) | Pre-Bolus and Post-Bolus (1hr, 3hr, 5hr)
Change in Fasting Glucose | Pre-Bolus and Post-Bolus (1hr, 3hr, 5hr)
Change in Systolic and Diastolic Blood Pressure | Pre-Bolus and Post-Bolus (30min, 1hr, 2hr, 3hr, 4hr, 5hr)

SECONDARY OUTCOMES:
Change in Augmentation Index | Pre-Bolus and Post-Bolus (30min, 1hr, 2hr, 3hr, 4hr, 5hr)
  Measure of arterial stiffness and central blood pressures
Change in Aortic Systolic and Diastolic Pressure | Pre-Bolus and Post-Bolus (30min, 1hr, 2hr, 3hr, 4hr, 5hr)
  Measure of arterial stiffness and central blood pressures
Change in Augmentation Pressure | Pre-Bolus and Post-Bolus (30min, 1hr, 2hr, 3hr, 4hr, 5hr)
  Measure of arterial stiffness and central blood pressures
Change in Cardiac Output | Pre-Bolus and Post-Bolus (30min, 1hr, 2hr, 3hr, 4hr, 5hr)
  Beat-to-beat resting cardiac haemodynamics (cardiac output, mean arterial pressure, strove volume, total peripheral resistance, heart rate)
Change in Stroke Volume | Pre-Bolus and Post-Bolus (30min, 1hr, 2hr, 3hr, 4hr, 5hr)
  Beat-to-beat resting cardiac haemodynamics
Change in Heart Rate | Pre-Bolus and Post-Bolus (30min, 1hr, 2hr, 3hr, 4hr, 5hr)
  Beat-to-beat resting cardiac haemodynamics
Change in Mean Arterial Pressure | Pre-Bolus and Post-Bolus (30min, 1hr, 2hr, 3hr, 4hr, 5hr)
  Beat-to-beat resting cardiac haemodynamics
Change in Total Peripheral Resistance | Pre-Bolus and Post-Bolus (30min, 1hr, 2hr, 3hr, 4hr, 5hr)
  Beat-to-beat resting cardiac haemodynamics
Change in Resting Energy Expenditure | Pre-Bolus and Post-Bolus (30min, 1hr, 2hr, 3hr, 4hr, 5hr)
  Measured from indirect calorimetry
Change in Respiratory Quotient | Pre-Bolus and Post-Bolus (30min, 1hr, 2hr, 3hr, 4hr, 5hr)
  Measured from indirect calorimetry

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hertfordshire, Hatfield, United Kingdom